CLINICAL TRIAL: NCT06628739
Title: Correlation Between Imatinib Trough Concentration and Efficacy in Advanced Gastrointestinal Stromal Tumors Patients with Different Genotypes
Brief Title: Correlation Between Imatinib Trough Concentration and Efficacy in Advanced GIST Patients with Different Genotypes
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xinhua Zhang, MD, Deputy Director, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: No.[2023]184
Record Dates: First submitted 2024-05-27; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Stromal Tumor, Malignant
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — plasma for imatinib steady-state trough concentration measuring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IM Cmin below deciles boundary: Patients with imatinib Cmin less than the decile boundary based on each imatinib Cmin distribution decile.
- IM Cmin above deciles boundary: Patients with imatinib Cmin greater than or equal to the decile boundary based on each imatinib Cmin distribution decile.

INTERVENTIONS:
Drug: Imatinib — The long-term maintenance dose of every patient was determined by the physician based on the guidelines and the patients' individual conditions such as adverse reactions.
  Other Names: Higher or lower imatinib Cmin

SUMMARY:
Imatinib (IM) has significantly enhanced the prognosis of patients (pts) with advanced gastrointestinal stromal tumors (GISTs). The clinical outcomes may correlate with IM exposure. However, the efficacy threshold, particularly based on different primary KIT mutant, remains undefined. The objective of this study is to establish the efficacy threshold of imatinib (IM) plasma trough concentration (Cmin) at steady-state in Chinese patients with advanced GIST, additionally to define subgroup thresholds based on various primary KIT mutations.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors (GISTs) are the most common mesenchymal tumors of the gastrointestinal tract. The majority of GIST are driven by activating mutuations of KIT (60-70%) or platelet-derived growth factor receptor alpha (PDGFRA, 10-15%), in which KIT exon 11 mutation (52-58%) and KIT exon 9 mutation (6-9%) are the most common types of KIT mutations. Patients with different activating KIT mutations have different sensitivity to imatinib therapy. In the first-line therapy, patients with KIT exon 11 mutation receiving Imatinib with standard dose of 400mg/d has the best therapeutic effect. Patients with KIT exon 9 mutation have poor sensitivity to the standard dose of imatinib, while higher doses can lead to better outcomes. The clinical outcomes may correlate with IM exposure. However, the efficacy threshold of imatinib in Chinese patients with advanced GIST remains unclear. The investigators aim to establish the efficacy threshold of imatinib plasma trough concentration (Cmin) at steady-state in Chinese patients with advanced GIST, additionally to define subgroup thresholds based on various primary KIT mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or recurrent GIST
* Aged 18 or older
* Treated with imatinib as first-line therapy
* Had imatinib Cmin measurement at steady state(at least one month after treatment) ≥2 times under long-term maintenance dose of regular medication
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2

Exclusion Criteria:

* Poor appliance
* Important treatment data missing
* Combined use of CYP enzyme inducers or inhibitors, such as rifampicin, carbamazepine, ketoconazole, ritonavir, rifamequal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From July 2017 to June 2022, 168 patients with advanced GIST who received imatinib treatment regularly and had pharmacokinetic (PK) blood samples availabe were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | through study completion, an average of 1 year
  Progression free survival (PFS) was defined as time from initiation of imatinib treatment until disease progression, as assessed by Choi criteria, or death caused by any reason.

SECONDARY OUTCOMES:
objective response rate | through study completion, an average of 1 year
  Objective response rate (ORR) was defined as rate of Complete Response (CR) and Partial Response (PR).
Overall survival | through study completion, an average of 1 year
  Overall survival (OS) was defined as time from initiation of imatinib treatment until death caused by any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xinhua, Professor, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No